CLINICAL TRIAL: NCT04235179
Title: Adjuvant Stereotactic Pelvic Irradiation in Endometrial Cancer (ASPIRE)
Brief Title: Adjuvant Stereotactic Pelvic Irradiation in Endometrial Cancer
Acronym: ASPIRE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Dr. Yasir Alayed, Consultant and Assistant Professor, King Saud University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E-19-4466
Record Dates: First submitted 2020-01-16; First posted 2020-01-21 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SABR (Experimental): Pelvic SABR for post-op endometrial cancer
  Interventions: Radiation: SABR

INTERVENTIONS:
Radiation: SABR — SABR to a dose of 30Gy/5 to the pelvis (vaginal and paravaginal tissues as well as regional lymph nodes)

SUMMARY:
Stereotactic Ablative Radiation (SABR/SBRT) will be prescribed to a dose of 30 Gy in 5 fractions, once weekly to the pelvis in post operative patients with endometrial cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patient with histologically confirmed endometrial adenocarcinoma
* Patient is a candidate for adjuvant pelvic radiation (+/- vault brachytherapy), meeting one of the following conditions: High grade histology OR Outer-half myometrial invasion with any risk factors OR FIGO stage II - IIIC1.
* Age ≥18 years.
* Patients who are to receive adjuvant systemic therapy in addition to pelvic radiotherapy will be eligible provided that there is at minimum a 3-week interval between any radiation treatment and chemotherapy treatments.

Exclusion Criteria:

* Patient has had prior pelvic radiotherapy.
* Patient has Type II endometrial cancer histology (ie. Serous, clear cell or carcinosarcoma).
* Patient has a contraindication to pelvic radiotherapy, such as but not limited to a connective tissue disease or inflammatory bowel disease.
* Patient has a contraindication to CT contrast.
* Patient has a hip prosthesis.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-01-16 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Acute Treatment-Related Adverse Events | 3 months after accrual is completed
  The number of participants with acute (<3 months) urinary and bowel treatment-related adverse events as assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0) criteria

SECONDARY OUTCOMES:
Late Treatment-Related Adverse Events | 5 years after accrual is completed
  The number of participants with late (>3 months) urinary and bowel treatment-related adverse events as assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0) criteria
Disease Local-Regional Failure Rate | 5 years after accrual is completed
  The rate of local-regional failure of the disease in participants after adjuvant SABR treatment in the setting of high-risk endometrial cancer.
Quality of Life | 5 years after accrual is completed
  The mean decrease in Quality of Life in participants after adjuvant SBRT treatment using EORTC (European Organisation for Research and Treatment of Cancer) core questionnaire (QLQ-C30) with EN-24 companion.

CONTACTS AND LOCATIONS:
Locations (1):
- King Saud University Medical City, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No